CLINICAL TRIAL: NCT06603025
Title: Investigation of the Effect of Preoperative Gum Chewing on Anxiety, Gastrointestinal Function, Nausea and Vomiting in Patients Undergoing Abdominal Surgery: a Randomized Controlled Trial
Brief Title: Preoperative Chewing Gum on Anxiety and Postoperative Nausea and Vomiting, Gastrointestinal Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülten Sucu Dağ, Assoc Prof Dr, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: GSD-2
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Gum Chewing; Preoperative; Anxiety; Postoperative Nausea and Vomiting
Keywords: Chewing Gum; Abdomen/surgery,; Postoperative Complications; Gastrointestinal Function; Ileus
MeSH Terms: conditions — Anxiety Disorders; Postoperative Nausea and Vomiting; Postoperative Complications; Ileus | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial with experimental and control groups
Who Masked: Outcomes Assessor
Masking Description: The statistician will not know which group the intervention is for. Data entry will be made as A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Preoperative intervention group patients will chew sugarless gum for at least 30 minutes 30-60 minutes before surgery. The gum will be removed before going to the operating room.
  Interventions: Other: chewing gum
- Control group (No Intervention): standard care (no chewing gum)

INTERVENTIONS:
Other: chewing gum — Preoperative intervention group patients will chew sugarless gum for at least 30 minutes 30-60 minutes before surgery. The gum will be removed before going to the operating room.
  Arms: Intervention group

SUMMARY:
The aim of this study was to investigate the effects of chewing gum before surgery on preoperative anxiety, postoperative gastrointestinal functions (time to first gas, time to first defecation, bowel sounds, abdominal distension) and nausea and vomiting in patients undergoing abdominal surgery.

Hypotheses of the Study: In patients undergoing abdominal surgery; H1.1: The first gas output time (hour) is shorter in patients who chew gum before surgery compared to patients who do not chew gum

H1.2: The first defecation time (hour) is shorter in patients who chew gum before surgery compared to patients who do not chew gum

H1.3: The bowel sounds are heard shorter in patients who chew gum before surgery compared to patients who do not chew gum H1.4: The abdominal distension rate is lower in patients who chew gum before surgery compared to patients who do not chew gum H1.5: The nausea and vomiting rate is lower in patients who chew gum before surgery compared to patients who do not chew gum H1.6: Preoperative anxiety levels of patients who chew gum before surgery are lower than those of patients who do not chew gum

Preoperative intervention group patients will chew sugarless gum for at least 30 minutes 30-60 minutes before surgery. The gum will be removed before going to the operating room. No intervention will be performed on control group patients, and standard care will be applied.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of chewing gum before surgery on preoperative anxiety, postoperative gastrointestinal functions (time to first gas, time to first defecation, bowel sounds, abdominal distension) and nausea and vomiting in patients undergoing abdominal surgery.

This study will be conducted as a single-center prospective randomized controlled trial in accordance with the principles of the Declaration of Helsinki. The study will be conducted in a private hospital in the Gazimağusa region on patients who will undergo abdominal surgery. Preoperative intervention group patients will chew sugarless gum for at least 30 minutes 30-60 minutes before surgery. The gum will be removed before going to the operating room. No intervention will be performed on control group patients, and standard care will be applied.

Sample inclusion criteria

* Patients with ASA scores I and II (ASA Physical Status Classification System)
* Patients with BMI < 30 (kg/m2)
* Patients over the age of 18 who will undergo abdominal surgery
* Patients who have the ability to read and understand the research instructions
* Patients who agree to participate in the research Sampling exclusion criteria
* Patients who do not accept chewing gum The number of samples to be included in the study was calculated by taking into account the median values of the first gas outlet time in the study of Bang et al. (2022). Accordingly, the median values of the first gas outlet time were 26.4 [15.2-39.2] hours in the control group and 20.6 [16.8-38.9] hours in the experimental group (Bang et al. 2022). Accordingly, it was planned to include a total of 70 patients, with an effect size of d = 0.70, a margin of error of α = 0.05, and a power of 80%, with a required sample size of 35 in each group. Considering that there may be missing data, it was decided to increase the sample size by 10% and include 39 patients in each group, making a total of 78 patients.

The time to first gas discharge after surgery, the time to first defecation, the duration of hospital stay, the frequency of nausea, vomiting and abdominal distension, the time and number of bowel sounds heard, and the need for antiemetic medication after surgery will be recorded in the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II
* body mass index (BMI) < 30 (kg/m2)
* individuals undergoing abdominal surgery

Exclusion Criteria:

* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
the preoperative anxiety | before entering OR
  the preoperative anxiety using APAIS immediately before entering OR. The APAIS scale consists of 6 items, and each statement is given a numerical value based on a 5-point Likert scale according to severity. These values, which vary between 1-5; 1=none, 2=mild, 3=moderate, 4=severe, 5=extremely severe. The scores on the anxiety of APAIS range from 6 (not anxious) to 30 (extremely anxious).

SECONDARY OUTCOMES:
abdominal distantion | 1 day after surgery. after surgery, the patient will be evaluated every 4 hours up to 48-72 hours after surgery
  abdominal distension (frequency). abdominal distantion will be evaluated by performing an abdominal examination every 4 hours. Abdominal distension will be evaluated as present or absent after the evaluation.
nausea, vomiting | 1 day after surgery. The patient will be asked every 4 hours whether they have nausea/vomiting up to 48-72 hours after surgery
  nausea and vomiting(frequency). The patient will be asked whether they have nausea/vomiting. The patients nausea and vomiting status and frequency will be recorded.
Time to first flatus | after surgery until the first flatus up to 48-72 hours
  The mean time to first flatus (hours). The time to first flatus will be evaluated by asking the patient after the surgery. If there is gas discharge, it will be evaluated as yes and the time of gas discharge after the surgery will be recorded.
Time to first bowel movement | after surgery until the first bowel movements up to 48-72 hours
  Time to first bowel sounds (Hours). Patients bowel movements will be examined abdominally using a stethoscope to detect the intestinal movement every 4 hours
first defecation time | after surgery until the patients defecation time up to 48-72 hours
  The mean time to first defecation time (hours). The time to first defecation time will be evaluated by asking the patient after the surgery. If there is first defecation, it will be evaluated as yes and the time of first defecation after the surgery will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, North Cyprus Via Mersin, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang YJ, Lee JH, Kim CS, Lee YY, Min JJ. Anxiolytic effects of chewing gum during preoperative fasting and patient-centered outcome in female patients undergoing elective gynecologic surgery: randomized controlled study. Sci Rep. 2022 Mar 9;12(1):4165. doi: 10.1038/s41598-022-07942-6. PMID 35264684
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8907183/